CLINICAL TRIAL: NCT02828436
Title: A Pilot Study to Assess Spinal Cord Stimulation To Inhibit Afferent Feedback During Exercise in Hypertension
Brief Title: Spinal Cord Stimulation to Treat Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1604M86961
Record Dates: First submitted 2016-06-15; First posted 2016-07-11 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Hypertension
Keywords: Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Spinal Cord Stimulation (Experimental): Boston Scientific Precision Spectra System
  Interventions: Device: Precision Spectra System
- Exercise Intervention (Other): If subject cannot tolerate Spinal Cord stimulation they will be assigned this arm
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Device: Precision Spectra System — Spinal Cord Stimulation
  Arms: Spinal Cord Stimulation
Behavioral: Exercise Intervention — Standard Exercise
  Arms: Exercise Intervention

SUMMARY:
To investigate the exercise blood pressure response during a lower-extremity dynamic exercise in postmenopausal women with hypertension and to determine if lumbar epidural spinal cord stimulation reduces blood pressure during exercise in postmenopausal women and men with hypertension.

DETAILED DESCRIPTION:
This is a single center study conducted at the University of Minnesota, enrolling up to forty subjects (30 men and 30 post-menopausal women). Subjects will be a assigned to one of the two study arms, (Dynamic Exercise or Spinal Cord Stimulation) and then crossover to the other arm after the initial assignment is complete. However is the screening MRI determines the subject is not a candidate for spinal cord stimulation, then they will be assigned to the Dynamic Exercise arm only.

ELIGIBILITY:
Inclusion Criteria:

1. Men and post-menopausal women between the ages of 40-90 years old
2. Hypertension (defined as BP ≥ 140/90), diagnosed by a physician
3. Ability of the patient to provide consent

Exclusion Criteria:

1. History of cardiopulmonary disorders other than hypertension, as determined on the medical evaluation questionnaire.
2. History of dangerous arrhythmias (arrhythmias requiring treatment or requiring physician supervision)
3. Currently taking specific anti-hypertensive medications that may affect the exercise pressor response or influence the effect of spinal cord stimulation.

   Please contact study staff for information regarding your eligibility.
4. History of spinal fusion or laminectomy at L3 or above
5. Current prescription opioid usage
6. Contraindication to MRI
7. At physician discretion which will be documented on the case report form.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manda Keller-Ross, PhD, DPT, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Spinal Cord Stimulation | Exercise Intervention
Started | 0 | 9
Completed | 0 | 5
Not Completed | 0 | 4
Not completed — Did Not Meet Inclusion Criteria | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Period: Period 2
Arm/Group | Spinal Cord Stimulation | Exercise Intervention
Started | 9 | 0
Completed | 1 | 0
Not Completed | 8 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Did Not Meet Inclusion Criteria | 3 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only participants who completed the study are included in the baseline analysis.
Groups:
- All Participants: This is a cross-over study. All participants are pooled at baseline.
Arm/Group | All Participants
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Pressor Reflex From Baseline
Description: Change in blood pressure during exercise.
Time Frame: 2 years
Measure: Mean (Standard Error); unit: mmHG
Arm/Group | Spinal Cord Stimulation | Exercise Intervention
Number analyzed (Participants) | 1 | 5
mmHG | 8.67 (NA) — Only one participant included in this arm. Standard error is not applicable. Data reported were collected during dynamic exercise arm. | 16.29 (1.82)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Spinal Cord Stimulation | Exercise Intervention
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 0/1 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT02828436/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT02828436/ICF_001.pdf